CLINICAL TRIAL: NCT04710810
Title: Transplantation of Human Allogenic Cord Blood Mononuclear Stem Cells in Autism: Safety and Efficacy of the Method
Brief Title: UCB Stem Cells for Autism Spectrum Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Petersburg Bekhterev Research Psychoneurological Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCA1512
Record Dates: First submitted 2020-12-28; First posted 2021-01-15 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients receive group and rhesus compatible UCB cells through intravenous bolus injections (4 injections at 2-week intervals) after pre-medication with Clemastine (0.025 mg/kg body weight, intravenously). One dose is 250±10 x 10⁶ viable cells per sample.
  Interventions: Other: umbilical cord blood mononuclear stem cells
- Control (No Intervention): Patients receives standard therapy (applied behavioral analysis, speech therapy).

INTERVENTIONS:
Other: umbilical cord blood mononuclear stem cells — UCB samples (70-130 ml of initial volume) were aseptically drained in blood-collection bags with 35 mL of citrate phosphate dextrose (CPDA-1) anticoagulant. Red blood cell-depleted/plasma-reduced nucleated cells were isolated by sedimentation in dextran-40, resuspended in autologous plasma with 10% dimethylsulfoxide and 1% dextran-40, and aliquoted in 3.8 ml vials with target doses of 3.0±0.2 x 10⁶ cells per vial. Vials were cooled to -90⁰C, quarantined in the vapor phase of liquid nitrogen. Tested for HIV-1/2, hepatitis B and C, HTLV-1/2, HSV-1 and -2, CMV, syphilis, and sterility. Characterized by AB0/Rh, CD34/CD45-positive cell content. Before injection sample thaws in the water bath at +37⁰C and washes from an excess amount of DMSO in 40 mL of physiological saline containing 2.5% human serum albumin and 5% dextran-40. After centrifugation and supernatant withdrawal, the UCB resuspends in 40 ml of the same solution at a target dose of 250±10 x 10⁶ viable cells per sample.
  Arms: Experimental

SUMMARY:
Purpose. The goals of the study are to assess the safety of the intravenous infusion of umbilical cord blood (UCB) cells in patients with autism and to confirm changes in social/ communicative skills and cognitive functioning after four infusions of ABO/Rh-matched UCB stem cells.

Material and methods. The sample comprises 30 patients (27 males, 3 females) aged between 3 and 11 years with ASD under the care of the National Medical Research Center for Psychiatry and Neurology (Saint-Petersburg, Russia). Participants are randomly assigned to either the control group (14 males, 1 female) or the experimental group (13 males, 2 females). The experimental group receives intravenous injections of UCB cells four times with a two-week gap between injections. The control group receives standard therapy.

The dynamic of cognitive functions and social/communicative skills assess with Checklist for autism spectrum disorders (CASD), Autism treatment evaluation checklist (ATEC), subscales of Wechsler Intelligence Scale for Children (WISC) - "Digit Span", "Picture completion", "Block design", "Coding".

ELIGIBILITY:
Inclusion Criteria:

* diagnosed ASD by ICD-10 criteria

Exclusion Criteria:

* acute somatic diseases
* indication for surgical (neurosurgical) therapy
* acute or chronic infectious diseases
* history of acute allergic reactions

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 24 hours after infusion
  Assessed by Adverse Event Grading Scale. It categorized adverse events according to severity.
  Mild Adverse Event - event results in mild or transient discomfort, not requiring intervention or treatment; does not limit or interfere with daily activities (e.g., insomnia, mild headache).
  Moderate Adverse Event - event is sufficiently discomforting so as to limit or interfere with daily activities; may require interventional treatment (e.g., fever requiring antipyretic medication).
  Severe and undesirable Adverse Event - event results in significant symptoms that prevent normal daily activities; may require hospitalization or invasive intervention (e.g., anemia resulting in blood transfusion).
Changes in severity of autistic symptoms from baseline at 3d and 6th month (measured by Checklist for Autism Spectrum Disorders (CASD) | at baseline, 3d and 6th month
  The CASD rates 30 symptoms of autism, covering six domains: problems with social interaction, perseveration, somatosensory disturbance, atypical communication and development, mood, problems with attention and safety. Symptoms are scored as present or absent based on information drawn from various sources, including teacher, caregiver, parent, observation of the child, and available records. The scores from each subscale are combined in order to calculate a Total Score, which ranges from 0 to 30 points. A lower score indicates less severe symptoms of ASD and a higher score correlates with more severe symptoms of ASD.
Changes in severity of autistic symptoms from baseline at 3d and 6th month (measured by Autism Treatment Evaluation Checklist (ATEC) | at baseline, 3d and 6th month
  The purpose of the ATEC is to measure a change in a patient due to various interventions. It consists of four subtests: Speech/Language Communication (14 items); Sociability (20 items); Sensory/ Cognitive Awareness (18 items); Health/Physical/Behavior (25 items). The scores from each subscale are combined in order to calculate a Total Score, which ranges from 0 to 179 points. A lower score indicates less severe symptoms of ASD and a higher score correlates with more severe symptoms of ASD.

SECONDARY OUTCOMES:
"Digit Span" subscale of Wechsler Intelligence Scale for Children (WISC) | at baseline, 6th month
  It assesses short-term auditory memory, concentration. The child is asked to repeat dictated series of digits forwards and other series backwards. Series begin with two digits and keep increasing in length, with two trials at each length. A primary score ranges from 0 to 9 points for forward series and from 0 to 8 points for backward series. The primary score is further converted into a final score in accordance with the age of the patient. A higher score correlates with better cognitive functioning.
"Picture completion" subscale of Wechsler Intelligence Scale for Children (WISC) | at baseline, 6th month
  This subscale measures alertness to detail, visual discrimination. The child is asked to identify missing parts of pictures. A primary score ranges from 0 to 20 points. The primary score is further converted into a final score in accordance with the age of the patient. A higher score means better cognitive functioning.
"Block design" subscale of Wechsler Intelligence Scale for Children (WISC) | at baseline, 6th month
  It helps to measure spatial analysis, abstract visual problem-solving. It provides blocks and pictures, and the child must put the blocks together to re-create what's in the picture of the blocks. A primary score ranges from 0 to 55 points. The primary score is further converted into a final score in accordance with the age of the patient. A higher score means better cognitive functioning.
"Coding" subscale of Wechsler Intelligence Scale for Children (WISC) | at baseline, 6th month
  It assesses visual-motor coordination, speed, concentration. Coding A is used for children under age 8. The child is asked to mark rows of shapes with different lines according to a code as quickly as possible for 2 minutes. A primary score ranges (Coding A) from 0 to 50 points. Coding B is used for children aged 8 and older. The child is asked to transcribe a digit-symbol code as quickly as possible for two minutes. A primary score ranges (Coding B) from 0 to 93 points. The primary score is further converted into the final score in accordance with the age of the patient. A higher score means better cognitive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- St.-Petersburg Bekhterev Reserach Psychoneurological Institute, Saint Petersburg, Sankt-Peterburg, Russia